CLINICAL TRIAL: NCT03180541
Title: Evaluation of a Coordinated National Implementation of DBT in Community Mental Health Services in Ireland
Brief Title: Evaluating the Coordinated National Implementation of DBT in Ireland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Service Executive, Ireland (Other)
Responsible Party: Principal Investigator, Mary Joyce, Project Co-ordinator, Health Service Executive, Ireland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOSP 2
Record Dates: First submitted 2017-05-24; First posted 2017-06-08 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Personality Disorder, Borderline
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialectical Behaviour Therapy (Experimental): Participants receive the "standard" 12 month DBT programme where all four modes of treatment are delivered including: individual therapy, group skills training, telephone coaching and DBT team consultation
  Interventions: Behavioral: Dialectical Behaviour Therapy
- Treatment-As-Usual (No Intervention): The Treatment-As-Usual arm will include individuals who:
  * live in areas where no DBT intervention is currently available OR
  * were offered a place on the DBT programme but decided not to partake at that time

INTERVENTIONS:
Behavioral: Dialectical Behaviour Therapy — Dialectical Behaviour Therapy (DBT) is a psychological intervention which was originally developed for women with Borderline Personality Disorder. DBT is delivered by a team of multidisciplinary mental health professionals, and comprises of individual therapy sessions for each patient, group skills training sessions, phone coaching and consultation meetings for the clinicians on the DBT team. Group skills are delivered in blocks of three modules which teach mindfulness, distress tolerance, emotion regulation and interpersonal effectiveness. The three modules are delivered over a 24-week period and are then repeated.
  Arms: Dialectical Behaviour Therapy

SUMMARY:
This study aims to evaluate the coordinated implementation of Dialectical Behaviour Therapy in Community Mental Health Services in Ireland.

There are three main objectives of the current study:

* evaluate the effectiveness of DBT for adults and adolescents attending Community Mental Health Services in multiple sites across Ireland
* conduct an economic evaluation of the coordinated implementation of DBT in community settings in Ireland
* evaluate the implementation initiative by means of quantity, quality and experience of the coordinated implementation

DETAILED DESCRIPTION:
The National Dialectical Behaviour Therapy (DBT) Project, Ireland was established in the Republic of Ireland in 2013. The aims of the project were twofold: to implement DBT in Community Mental Health Services across Ireland and to evaluate this coordinated implementation of DBT at a national level.

DBT was initially formulated as a treatment for Borderline Personality Disorder (BPD) which is typically characterised by patterns of emotional and behavioural dysregulation that often manifests in self-harm and suicidal ideation. DBT is noted to be an intervention with a growing evidence base that demonstrates its effectiveness in treating individuals with BPD. More than a dozen controlled trials have been completed at multiple independent sites. The results of these trials have reported a reduction in suicidal behaviours, inpatient hospitalisations, depression, hopelessness and suicidal ideation among other constructs which individuals with BPD experience.

While the efficacy of DBT has been demonstrated through multiple controlled trials, few studies have examined the effectiveness of DBT in community mental health settings. In particular, no study has evaluated a coordinated national implementation of DBT across multiple sites in a publicly funded health system. The current study aims to evaluate the the coordinated implementation of DBT in Community Mental Health Services in Ireland

ELIGIBILITY:
Inclusion Criteria:

Adults:

* Meet criteria for diagnosis of either Borderline Personality Disorder (DSM IV/V) or Emotionally Unstable Personality Disorder (ICD-10)
* A persistent pattern of deliberate self-harm with deliberate self-harm behaviour having occurred within the last 6 months OR one suicidal act having occurred within the last 6 months
* The individual will have discussed the diagnosis with a member of the DBT team and will have expressed an interest in, and commitment to the 12 month programme.

Adolescents:

* Between/ including the ages of 13 and 18 years
* Demonstrating emotional behavioural disturbance/ emotional dysregulation
* A persistent pattern of deliberate self-harm with deliberate self-harm or a suicidal act having occurred within the last 16 weeks OR chronic suicidal ideation
* the young person and their parent/guardian will have discussed their emotional behavioural disturbance/ emotional dysregulation with a member of the DBT team and will have expressed an interest in, and commitment to the 16 week programme.

Exclusion Criteria:

Adults and Adolescents:

* An active psychosis
* If the client has severe developmental delays, cognitive impairment or learning disabilities (exceeding mild range)
* If a clients' substance/drug dependence, eating disorder or any other mental health issue/behaviour is at such a level that it would impede their engaging with any of the modalities of DBT

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in self-harm behaviour | Pre-intervention, 6 months, 12 months (post-intervention) and 18 months (6 months post-intervention)
  Change in frequency of self-harm behaviour. Frequency of self-harm behaviour for a six month period will be recorded by the DBT therapist working with each individual by means of clinical file review. Self-harm behaviour frequency is scored on a scale of 1 to 5 where 1 = Not at all, 2 = Rarely; 3 = Occasionally, 4 = Often, 5 = Most of the time.
Change in borderline symptoms | Pre-intervention, 6 months, 12 months (post-intervention) and 18 months (6 months post-intervention)
  Borderline Symptom List (BSL-23). The BSL-23 is a self-report questionnaire which comprises 23 items measuring borderline-typical symptomatology.
Change in suicidal ideation | Pre-intervention, 6 months, 12 months (post-intervention) and 18 months (6 months post-intervention)
  Questionnaire for Suicidal Ideation (QSI). The QSI is a 6-item self-report questionnaire developed by the researchers to assess suicidal thoughts and ideation.

SECONDARY OUTCOMES:
Change in depression | Pre-intervention, 6 months, 12 months (post-intervention) and 18 months (6 months post-intervention)
  Beck Depression Inventory - Second Edition (BDI-II). The BDI-II is a 21 item self-report measure of symptoms and attitudes related to depression.
Change in hopelessness | Pre-intervention, 6 months, 12 months (post-intervention) and 18 months (6 months post-intervention)
  Beck Hopelessness Scale (BHS). The BHS is a 20 item self-report measure which assesses key aspects of hopelessness.
Change in DBT Skill Use | Pre-intervention, 6 months, 12 months (post-intervention) and 18 months (6 months post-intervention)
  DBT Ways of Coping Checklist (DBT-WCCL). The DBT-WCCL is a 59-item self-report measure which assesses DBT skill use and dysfunctional coping.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Flynn, Prof. Dip, Principal Investigator — Psychology Manager

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flynn D, Joyce M, Gillespie C, Kells M, Swales M, Spillane A, Hurley J, Hayes A, Gallagher E, Arensman E, Weihrauch M. Evaluating the national multisite implementation of dialectical behaviour therapy in a community setting: a mixed methods approach. BMC Psychiatry. 2020 May 14;20(1):235. doi: 10.1186/s12888-020-02610-3. PMID 32410670
- [Derived] Flynn D, Kells M, Joyce M, Suarez C, Gillespie C. Dialectical behaviour therapy for treating adults and adolescents with emotional and behavioural dysregulation: study protocol of a coordinated implementation in a publicly funded health service. BMC Psychiatry. 2018 Feb 26;18(1):51. doi: 10.1186/s12888-018-1627-9. PMID 29482538